CLINICAL TRIAL: NCT07336784
Title: Impact of Simulation-Based Teaching on Knowledge Acquisition in Anesthesiology Residents During Wartime: A Randomized Pilot Trial
Brief Title: Impact of Simulation-Based Teaching on Knowledge Acquisition in Anesthesiology Residents During Wartime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Institute, Ministry of Health of Ukraine (Other)
Collaborators: PL Shupyk National Healthcare University of Ukraine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: UA00000002025
Record Dates: First submitted 2025-12-18; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Medical Education; Anesthesiology Residency Training; Simulation-based Learning; Online Medical Education
Keywords: Simulation-based education; Simulation-based lectures; Online medical education; Anesthesiology residency training; Anesthesiology education; Medical education research; Randomized educational trial; Postgraduate medical education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation group (Experimental): Participants assigned to this arm received simulation-based lectures as part of the first-year anesthesiology residency curriculum. The intervention consisted of five simulation-based lectures, one for each educational component of the curriculum, delivered over a 3-month training period. Each simulation-based lecture included interactive, high-fidelity simulation scenarios designed to replicate real clinical situations in anesthesiology and intensive care, such as emergency resuscitation, acute cardiovascular conditions, and anesthesia-related complications. Residents actively participated in scenario-based decision-making, followed by structured debriefing sessions and theoretical discussions aligned with current clinical guidelines and protocols. Training was conducted using specialized simulators or high-fidelity patient manikins. All sessions were led by the same experienced faculty instructor.
  Interventions: Other: Simulation-based lectures
- Online group (No Intervention): Participants assigned to this arm received online lectures covering the same educational components and learning objectives as the simulation group. The intervention consisted of five online lectures, one for each educational component of the curriculum, delivered over the same 3-month training period. Online lectures were conducted via a web-based video conferencing platform and included didactic presentations, demonstrations of clinical cases, and interactive question-and-answer sessions. Residents were able to participate in real time, ask questions, and engage in discussions with the instructor and peers. All online lectures were delivered by the same faculty instructor to ensure consistency of educational content across study arms.

INTERVENTIONS:
Other: Simulation-based lectures — Simulation-based lectures were conducted using interactive scenarios that replicated real clinical situations, in which anesthesiology residents not only applied practical skills to make decisions under realistic conditions but also subsequently reviewed the theoretical foundations of the presented topics. This instructional approach involved the use of specialized simulators or high-fidelity patient models, allowing the recreation of various clinical states such as emergency resuscitation, acute heart failure, and anesthesia-related complications. During the subsequent theoretical presentation, residents received detailed theoretical information and feedback from instructors.
  Arms: Simulation group

SUMMARY:
The goal of this study is to learn whether simulation-based lectures are more effective than online lectures in improving knowledge acquisition and retention among first-year anesthesiology residents. The study also examines residents' satisfaction with the different teaching formats.

The main questions this study aims to answer are:

Do simulation-based lectures improve residents' knowledge more than online lectures one month after training? Do residents who participate in simulation-based lectures report higher satisfaction and better understanding of the material compared to those attending online lectures? Researchers will compare simulation-based lectures with online lectures covering the same educational topics to determine which teaching method is more effective for anesthesiology training.

Participants will:

Be randomly assigned to receive either simulation-based lectures or online lectures Attend five lectures (one per educational component) over a 3-month training period Complete a knowledge test before the lectures and again one month after the training Complete a final examination at the end of the curriculum Fill out a questionnaire evaluating their satisfaction with the training format

DETAILED DESCRIPTION:
This study is a randomized, prospective, pilot educational trial designed to compare the effectiveness of simulation-based lectures versus online lectures on knowledge acquisition, knowledge retention, and learner satisfaction among first-year residents in the specialty of Anesthesiology and Intensive Care.

The study was conducted at the P.L. Shupyk National Healthcare University of Ukraine during an active wartime period, which imposed significant limitations on traditional clinical training and access to in-person educational resources. The intervention was implemented as part of the standard first-year residency curriculum.

Participants were first-year anesthesiology residents enrolled in a 3-month educational program consisting of 540 total training hours. Residents were randomly assigned in a 1:1 ratio to one of two educational modalities:

1. simulation-based lectures or
2. online lectures. Randomization was performed using a computer-generated block randomization sequence with variable block sizes. Participation in the study was voluntary, and residents who declined participation were excluded from the analysis.

Both groups received lectures covering identical educational components and learning objectives. The simulation-based lecture group participated in interactive sessions using high-fidelity simulation scenarios designed to replicate real-life anesthesiology and intensive care situations. Each simulation session included scenario execution, structured debriefing, and a subsequent theoretical discussion aligned with current clinical guidelines. The online lecture group received the same educational content delivered via a web-based video conferencing platform, including case-based discussions and interactive question-and-answer segments.

Educational effectiveness was evaluated using a modified Kirkpatrick model (Levels 1 and 2). Knowledge acquisition and retention were assessed using a standardized multiple-choice test administered before the intervention and one month after completion of the lectures. Additional assessment included a summative final examination conducted at the end of the 3-month curriculum. Learner satisfaction and perceived usefulness of the educational format were evaluated using a structured questionnaire with Likert-scale and open-ended items.

This study did not involve therapeutic, diagnostic, or preventive medical interventions and did not affect patient care. All study procedures were limited to educational activities and assessments. Ethical approval was obtained from the appropriate institutional ethics committee, and written informed consent was obtained from all participants prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* First-year residents enrolled in the specialty of Anesthesiology and Intensive Care
* Enrollment in the first year of residency training at the Department of Anesthesiology and Intensive Care, P.L. Shupyk National Healthcare University of Ukraine
* Participation in the standard first-year residency curriculum during the study period
* Ability and willingness to provide written informed consent to participate in the study

Exclusion Criteria:

* Refusal to participate in the study
* Failure to complete the full training program (e.g., due to early termination of training, relocation abroad, or academic leave)
* Withdrawal from the study before completion of outcome assessments

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Knowledge Retention at 1 Month | 1 month after completion of the lectures
  Knowledge retention assessed one month after completion of the educational intervention using a standardized 15-item multiple-choice test covering five educational components of anesthesiology training. Each correct answer was awarded one point. Score range: 0-15 points, where higher scores indicate better knowledge acquisition, with 15 representing the best possible result.

SECONDARY OUTCOMES:
Immediate Knowledge Acquisition | Before the intervention
  Baseline knowledge level assessed before the educational intervention using the same standardized 15-item multiple-choice test. Each correct answer was awarded one point. Score range: 0-15 points, where higher scores indicate better knowledge acquisition, with 15 representing the best possible result.
Final Summative Examination Performance | End of the 3-month training program
  Overall knowledge performance assessed at the end of the 3-month curriculum using a 30-item multiple-choice final examination covering all five educational components. Score range: 0-30 points, where higher scores indicate better result, with 30 representing the best possible result
Learner Satisfaction | End of the 3-month training program
  Participants' satisfaction was assessed using a structured questionnaire based on the Kirkpatrick Level 1 Evaluation Model (Reaction Level). The questionnaire included Likert-scale items with scores ranging from 1 to 5, where 1 = strongly disagree and 5 = strongly agree. The minimum possible score was 1 and the maximum possible score was 5. Higher scores indicate greater satisfaction and a better educational outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- PL Shupyk National Healthcare University of Ukraine, Kyiv, Kyiv Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this study may be shared upon reasonable request, subject to approval by the study investigators and the institutional ethics committee. Data will be shared for academic research purposes only, in accordance with applicable regulations and institutional policies.
Supporting Information: Study Protocol